CLINICAL TRIAL: NCT05917171
Title: Developing a Culturally Appropriate Non-Opioid Pain Coping Skills Training Intervention for Spanish-Speaking Patients With Cancer Pain Using a Community Engaged Approach
Brief Title: Pilot Trial of an Online Pain Coping Skills Training Program in Spanish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00096781
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-04

CONDITIONS: Cancer Pain
Keywords: pain coping skills; cancer-related pain; pain management
MeSH Terms: conditions — Cancer Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Single group pilot study to assess feasibility and acceptability.
Masking Description: Non-random pilot trial with no masking due to single group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- painTRAINER intervention (Experimental): 40 Spanish speaking Hispanic and Latine participants will participate in an 8 week online pain coping skills training program designed to address cancer-related pain.
  Interventions: Behavioral: painTRAINER

INTERVENTIONS:
Behavioral: painTRAINER — painTRAINER is an 8 week online behavioral pain coping skills training program derived from cognitive behavioral therapy approaches, which includes 45 minute behavioral coping sessions to be completed over 8 weeks. Weekly sessions are guided by an automated coach that teaches skills for coping with pain.

SUMMARY:
The goal of this pilot study is to assess the feasibility and acceptability of an 8-week online pain coping skills training program designed specifically for Spanish-speaking Hispanic and Latine populations experiencing cancer-related pain. The main questions aim to answer are: 1. what is the feasibility of this program for engaging and recruiting Spanish speaking members of the Hispanic and Latine community?; 2. How well is the program accepted by Spanish speaking members of the Hispanic and Latine community?. Participants will answer questions about their cancer related pain before and after they participate in an 8-week pain coping skills training program offered online.

DETAILED DESCRIPTION:
Cancer-related pain is a significant adverse effect of cancer and cancer treatment, which poses significant management challenges for patients. Compared to non-Hispanic whites, Spanish-speaking Hispanic patients routinely experience disparities in cancer-related care that negatively impact quality of life, including more significant barriers in accessing quality care, less adequate pain management, and later-stage cancer diagnosis and treatment initiation. Limited English proficiency is a particularly difficult barrier among primarily Spanish-speaking Hispanic patients, as communication challenges with providers contributes to poorer pain outcomes and suboptimal pain management. To support Spanish-speaking populations and strive towards more equitable care (e.g., accessible, convenient, and cost-effective), this study is leveraging its prior work in Pain Coping Skills Training (PCST) through the cultural and linguistic translation of an online PCST program, painTRAINER. This evidence-based program, delivered online over eight weeks, facilitates development of pain coping skills to improve pain outcomes while also reducing reliance on opioids for pain management.

This pilot study follows a community-engaged and community-driven approach for translating and adapting the painTRAINER program into a linguistically and culturally appropriate version optimized for diverse Spanish-speaking adults experiencing cancer-related pain.

The study team integrated Spanish-speaking staff, community members, community-based organizations, and key stakeholders as members of the research team to guide the program adaptation process. Community partners include key members of the Hispanic community and leaders from various community organizations, who have participated on the study's Community Advisory Board (CAB) and on a Community-based Programmatic Review Panel (PRP). Both groups include members from diverse Spanish speaking countries with diversity in age, gender, and educational background and have been integral in guiding the translation and adaptation process. This group continue to play a key role in future phases of the project such as participant recruitment, implementation, data analysis and interpretation, and dissemination of findings.

Prior studies show that PCST is effective, engaging, and acceptable to English-speaking patients, and also is an accessible, convenient, and cost-effective pain management tool when delivered online. PainTRAINER's effectiveness for pain management is well established via NIH-funded trials. Results from previous studies show critical implications in the development and delivery of pain management for underserved cancer populations to foster equity in care and reduce reliance on opioid medications. The community-engaged and culturally-informed process to fully adapt and translate the painTRAINER program will yield an effective Spanish-language PCST program that fills a gap in cancer-pain management by further expanding access to quality care among Hispanic patients. Community partnerships are key to the successful adaptation and future intervention efforts of the Spanish-language version of painTRAINER. The availability of effective and culturally-appropriate pain management options for Spanish-speaking patients will provide communities with tools and resources necessary not only for managing pain and enhancing quality of life, but for empowering Spanish-speaking patients to be strong advocates for their health.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive cancer treated with either single modality therapy or any combination of therapies.
* Is ≤ 5 years since completion of definitive cancer therapy.
* May be off treatment, receiving adjuvant or maintenance therapy or have cancer that is stable/controlled.
* Pain score ≥ 4 (PROMIS Pain Intensity (1a) scale) on "Most Days" or more (Graded Chronic Pain Scale).
* Pain of new onset or significantly exacerbated since cancer diagnosis or initiation of cancer treatment.
* If taking analgesics, the analgesic regimen must be stable; unexpected dose adjustments are allowed.
* Expected capable of completing study activities (clinician judgment) with ECOG performance status ≤ 2.
* Age ≥18 years at the time of study entry.
* Identify as Hispanic or Latine AND able to read and speak Spanish.

Exclusion Criteria:

* Has a disability that precludes completion of study activities.
* Reports only preexisting pain conditions unrelated to cancer or cancer treatment.
* Has a known or suspected diagnosable substance use disorder or opioid overuse disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Adherence - percent of participants who complete the study modules as a measure of retention | baseline
  To evaluate the feasibility of implementing painTRAINER among Spanish speaking participants, the study will assess participants' adherence to painTRAINER and the capacity to retain them in a clinical trial. The pilot trial can be implemented completely remotely among community dwelling Spanish-speaking Hispanic/Latine individuals with cancer-related pain. The study will calculate the percent of participants who complete the study modules as a measure of retention. Adherence to the program will be defined as the proportion of weekly modules completed (adequate adherence is defined as completion of ≥ 75% of modules, or 6 of the total 8 modules).
Adherence - percent of participants who complete the study modules as a measure of retention | Week 10
  To evaluate the feasibility of implementing painTRAINER among Spanish speaking participants, the study will assess participants' adherence to painTRAINER and the capacity to retain them in a clinical trial. The pilot trial can be implemented completely remotely among community dwelling Spanish-speaking Hispanic/Latine individuals with cancer-related pain. The study will calculate the percent of participants who complete the study modules as a measure of retention. Adherence to the program will be defined as the proportion of weekly modules completed (adequate adherence is defined as completion of ≥ 75% of modules, or 6 of the total 8 modules).
Adherence - percent of participants who complete the study modules as a measure of retention | Week 18
  To evaluate the feasibility of implementing painTRAINER among Spanish speaking participants, the study will assess participants' adherence to painTRAINER and the capacity to retain them in a clinical trial. The pilot trial can be implemented completely remotely among community dwelling Spanish-speaking Hispanic/Latine individuals with cancer-related pain. The study will calculate the percent of participants who complete the study modules as a measure of retention. Adherence to the program will be defined as the proportion of weekly modules completed (adequate adherence is defined as completion of ≥ 75% of modules, or 6 of the total 8 modules).
Acceptability - proportion of eligible participants screened and the proportion of eligible participants who consent to participate | Baseline
  To assess the acceptability of painTRAINER among Spanish speaking participants, the study will determine the ability to recruit participants into the pilot trial via networks of community partners in the Atrium Health: Wake Forest Baptist catchment area. To characterize our ability to recruit participants, the study will estimate the proportion of eligible participants screened and the proportion of eligible participants who consent to participate. The study also will closely monitor the rate of referrals to the program by providers. Acceptability of the program also will be assessed more subjectively via interviews with participants following completion of or termination from the pilot trial.
Acceptability - proportion of eligible participants screened and the proportion of eligible participants who consent to participate | Week 10
  To assess the acceptability of painTRAINER among Spanish speaking participants, the study will determine the ability to recruit participants into the pilot trial via networks of community partners in the Atrium Health: Wake Forest Baptist catchment area. To characterize our ability to recruit participants, the study will estimate the proportion of eligible participants screened and the proportion of eligible participants who consent to participate. The study also will closely monitor the rate of referrals to the program by providers. Acceptability of the program also will be assessed more subjectively via interviews with participants following completion of or termination from the pilot trial.
Acceptability - proportion of eligible participants screened and the proportion of eligible participants who consent to participate | Week 18
  To assess the acceptability of painTRAINER among Spanish speaking participants, the study will determine the ability to recruit participants into the pilot trial via networks of community partners in the Atrium Health: Wake Forest Baptist catchment area. To characterize our ability to recruit participants, the study will estimate the proportion of eligible participants screened and the proportion of eligible participants who consent to participate. The study also will closely monitor the rate of referrals to the program by providers. Acceptability of the program also will be assessed more subjectively via interviews with participants following completion of or termination from the pilot trial.

SECONDARY OUTCOMES:
Change in Pain interference scores | baseline, 10 weeks, 18 weeks
  To determine the preliminary efficacy of painTRAINER as an intervention for pain management, the study will assess whether painTRAINER yields significant improvements in the pain interference (measured by the Brief Pain Inventory) from baseline to the post-intervention assessments for Spanish-speaking cancer survivors with persistent cancer-related pain. Scores are rated via Likert scale for low to high interference.
Change in Pain severity scores | baseline, 10 weeks, 18 weeks
  To determine the preliminary efficacy of painTRAINER as an intervention for pain management, we will assess whether painTRAINER yields significant improvements in pain severity (as measured by the Brief Pain Inventory (BPI)) from baseline to the post-intervention assessments for Spanish-speaking cancer survivors with persistent cancer-related pain. Scores are rated via Likert scale for low to high pain severity.
Change in Fatigue scores | baseline, 10 weeks, 18 weeks
  Fatigue will be assessed via the PROMIS Fatigue questionnaire. Scores are rated via Likert scale for low to high fatigue.
Change in Sleep disturbance scores | baseline, 10 weeks, 18 weeks
  Sleep disturbance will be assessed via the PROMIS Sleep Disturbance questionnaire. Scores are rated via Likert scale for low to high sleep disturbance.
Change in Pain resilience scores | baseline, 10 weeks, 18 weeks
  Pain resilience will be assessed via the PROMIS Pain Resilience Scale. Scores are rated via Likert scale for low to high pain resilience.
Change in Cognitive Function scores | baseline, 10 weeks, 18 weeks
  Cognitive function will be assessed via the PROMIS Cognitive Function scale. Scores are rated via Likert scale for low to high cognitive function.
Change in Physical Function scores | baseline, 10 weeks, 18 weeks
  Physical function will be assessed via the PROMIS Physical Function scale. Scores are rated via Likert scale for low to high physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Penzien, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05917171/ICF_000.pdf